CLINICAL TRIAL: NCT05250830
Title: Non-invasive bioELEctroniC Treatment foR pOst-cesarean paiN (ELECTRON)
Brief Title: TrueRelief Efficacy for Post-cesarean Pain (ELECTRON)
Acronym: ELECTRON
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: TrueRelief, LLC (Industry)
Responsible Party: Principal Investigator, Kara M Rood, MD, Assistant Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2022H0046
Record Dates: First submitted 2022-01-25; First posted 2022-02-22 (Actual); Results first posted 2024-06-06 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-05

CONDITIONS: Post-cesarean Pain
Keywords: Post-cesarean pain; Non-opioid; Non-invasive device

STUDY DESIGN:
Intervention Model Description: Double blind, randomized, sham-controlled trial parallel arm study using TrueRelief as the experimental treatment and a TrueRelief device with sham capabilities as a placebo.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- TrueRelief device (Experimental): Patients receive an experimental procedure using a TrueRelief device.
  Interventions: Device: TrueRelief device
- Sham TrueRelief device (Sham Comparator): Patients receive a placebo procedure using a sham TrueRelief device that looks and operates identically to the experimental TrueRelief device but will not emit any high frequency current.
  Interventions: Device: Sham TrueRelief device

INTERVENTIONS:
Device: TrueRelief device — TrueRelief is an FDA-cleared treatment for chronic intractable pain, and as an adjunctive procedure in the management of post-surgical and post-traumatic acute pain. This 20,000 Hz high frequency electrical procedure is provided by clinicians trained in the use of the device and delivered via handheld steel-tipped probes to the source of pain and where pain is experienced.
  Arms: TrueRelief device
Device: Sham TrueRelief device — The placebo device looks and operates identically to the experimental TrueRelief device but will not emit any high frequency current.
  Arms: Sham TrueRelief device

SUMMARY:
This is a randomized trial of 134 individualized post-cesarean delivery who will be randomized to twice daily use of non-invasive bioelectronic treatment with TrueRelief device or identical appearing sham device for post-cesarean pain management.

ELIGIBILITY:
Inclusion Criteria:

• Post cesarean delivery (combined vaginal/cesarean deliveries are not eligible) Singleton, or twin gestation

Exclusion Criteria:

* Known history of opioid use disorder, by medical record review
* Contraindication to opioids
* Contraindications to both acetaminophen and ibuprofen
* Significant surgical procedures (e.g., hysterectomy) prior to randomization as pain trajectory will be completely different
* Fetal or neonatal death prior to randomization
* Inability to randomize on postoperative day 0
* Inability to participate in twice daily use of non-invasive bioelectronic treatment during inpatient stay as assessed by research staff
* Language barrier (non-English or Spanish speaking)
* Participation in another intervention study that influences the primary outcome in this trial

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 134 (Actual)
Dates: Start 2022-04-18 (Actual); Primary Completion 2023-03-16 (Actual); Study Completion 2023-04-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio State University Wexner Medical Center OB/GYN Maternal and Fetal Medicine, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TrueRelief Device | Sham TrueRelief Device
Started | 67 | 67
Completed | 67 | 66
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TrueRelief Device | Sham TrueRelief Device | Total
Number analyzed (Participants) | 67 | 67 | 134
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 67 | 67 | 134
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.5 (4.9) | 31.4 (4.8) | 30.95 (4.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 67 | 134
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 67 | 67 | 134

OUTCOME MEASURES:

1. Primary Outcome: Median of Total Inpatient Oral Opioids Consumption (in Morphine Milligram Equivalents) in Treatment With TrueRelief Device Versus Sham Comparator Groups.
Description: The primary outcome is the total postoperative opioid intake through hospital discharge. All opioid doses were converted to equianalgesic doses of morphine sulfate MME using standard ratios.
Time Frame: For primary day of cesarean to day of discharge (3 days)
Measure: Median (Inter-Quartile Range); unit: Morphine milligram equivalents
Arm/Group | TrueRelief Device | Sham TrueRelief Device
Number analyzed (Participants) | 67 | 66
Morphine milligram equivalents | 19.75 [0 to 52.50] | 37.50 [7.50 to 67.50]

2. Secondary Outcome: Number of Participants Who Received Opioid Refill Prescription in Non-invasive Bioelectronic Treatment With TrueRelief Device Versus Sham Comparator Groups After Discharge.
Description: Additional opioid prescriptions within 6 weeks postpartum in non-invasive bioelectronic treatment with TrueRelief device versus sham comparator to see the effect in decreasing the number of opioid refill prescriptions.
Time Frame: After discharge through study completion, an average of six weeks
Measure: Count of Participants; unit: Participants
Arm/Group | TrueRelief Device | Sham TrueRelief Device
Number analyzed (Participants) | 67 | 66
Participants | 1 | 7

3. Secondary Outcome: Morphine Milligram Equivalents (MME) Opioid Tablets Prescribed at Discharge in Non-invasive Bioelectronic Treatment With TrueRelief Device Versus Sham Comparator Groups.
Description: Oral opioid prescribed at discharge as Morphine milligram equivalents (MME) in non-invasive bioelectronic treatment with TrueRelief device versus sham comparator.
Time Frame: At the discharge up to 24 hours
Measure: Median (Inter-Quartile Range); unit: Morphine milligram equivalents
Arm/Group | TrueRelief Device | Sham TrueRelief Device
Number analyzed (Participants) | 67 | 66
Morphine milligram equivalents | 82.50 [0 to 90.00] | 90.00 [75.00 to 90.00]

4. Secondary Outcome: Number of Participants With Pain Scores of Greater Than 4 (BPI Score >4) at Discharge.
Description: The Brief Pain Inventory (BPI) includes self-assessment of pain scores in the previous 24 hours using a numerical scale from 0 to 10, with 0 representing no pain and 10 the worst pain imaginable. Moderate to severe pain (BPI score >4) in past 24 h,
Time Frame: At the discharge up to 24 hours.
Measure: Count of Participants; unit: Participants
Arm/Group | TrueRelief Device | Sham TrueRelief Device
Number analyzed (Participants) | 67 | 66
Participants | 57 | 61

5. Secondary Outcome: Rate of Wound Infection or Separation in Non-invasive Bioelectronic Treatment With TrueRelief Device Versus Sham Comparator Groups.
Description: Rate of wound infection or separation in non-invasive bioelectronic treatment with TrueRelief device versus sham comparator groups.
Time Frame: After cesarean delivery until six weeks postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | TrueRelief Device | Sham TrueRelief Device
Number analyzed (Participants) | 67 | 66
Participants | 0 | 2

6. Secondary Outcome: Breastfeeding Rates in Non-invasive Bioelectronic Treatment With TrueRelief Device Versus Sham Comparator Groups.
Time Frame: At hospital discharge
Measure: Count of Participants; unit: Participants
Arm/Group | TrueRelief Device | Sham TrueRelief Device
Number analyzed (Participants) | 67 | 66
Participants | 59 | 57

ADVERSE EVENTS:
Time Frame: From the day of cesarean until six weeks postpartum
Arm/Group | TrueRelief Device | Sham TrueRelief Device
All-Cause Mortality (participants affected / at risk) | 0/67 | 0/67
Serious Adverse Events (participants affected / at risk) | 0/67 | 0/67
Other Adverse Events (participants affected / at risk) | 0/67 | 0/67

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-20): https://cdn.clinicaltrials.gov/large-docs/30/NCT05250830/Prot_SAP_000.pdf